CLINICAL TRIAL: NCT03530540
Title: A Prospective Randomized Double Blinded Placebo Controlled Clinical Trial Evaluating the Combined Effect of Low-Intensity Extracorporeal Shockwave Therapy (LI-ESWT) and Vacuum Erectile Device Combined With Manipulation Exercises on Peyronies Disease.
Brief Title: Low-Intensity Extracorporeal Shockwave Therapy and Vacuum Erectile Device as a Treatment for Peyronies Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lund,MD, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20170201
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Active shockwaves
  Interventions: Device: low-intensity extracorporeal shockwave therapy; Device: Penile pump
- Placebo (Placebo Comparator): Placebo shockwaves
  Interventions: Device: Placebo LI-ESWT; Device: Penile pump

INTERVENTIONS:
Device: low-intensity extracorporeal shockwave therapy — Active shockwaves
  Arms: Intervention
Device: Placebo LI-ESWT — Placebo shockwaves
  Arms: Placebo
Device: Penile pump — both groups will be treated with a penile pump

SUMMARY:
Aim The primary aim is to examine whether LI-ESWT and vacuum erectile device (VED) followed by manipulation exercises has beneficial effect on PD patients compared to a placebo group.

Primary Outcome

* Peyronie's Disease Questionnaire (PDQ)
* Visual Analogue Scale score (VAS)
* International Index of Erectile Function 5 (IEFF-5)
* Penile curve measurements (gold standard) on pictures before and after treatment
* Plaque size

Method This study is designed as a prospective, randomized, double-blinded, placebo-controlled with follow-up after 1, 3 and 6 months.

A total of 50 participants who meets the inclusion criteria's will randomly be assigned to I(intervention) or C(control) group based on a randomization list which is retained in a sealed envelope. The content of the envelope is only familiar to the Head of the Department of Urology to ensure valid randomization.

All treatment sessions are executed at the outpatient clinic of the department of urology department L at Odense University Hospital(OUH). All patients receive treatment with the same device a Duolith® SD1 T-Top from Storz Medical. However, when treating patients in the control group the handpiece will be covered by a shockwave absorbent material. Settings and setup are identical in both groups to make sure that patients are unable to acknowledge which treatment is being performed.

ELIGIBILITY:
Inclusion Criteria:

* PD for more than 6 months
* Penile curve greater than 30 degrees and less than 90 degrees
* Age 18-80
* No previous penile surgery
* Informed consent
* Able to speak and understand Danish

Exclusion Criteria:

* Penile curve greater than 90 degrees
* Previous surgery for PD
* Patients undergoing other interventions for PD

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in penile curvature | penile curve will be assessed at baseline, and 1,3 and 6 months.
  Change in penile curvature from baseline to follow-up at 1,3 and 6 months. Penile curvature is measured on pictures submitted by the patient.

SECONDARY OUTCOMES:
Change in pain score using the Visual Analogue Scale (VAS) | VAS will be assessed at baseline, and 1,3 and 6 months.
  VAS is a subjective pain score ranging from 0-10 whereas 0 means no pain, and 10 being excruciating pain. Patients are asked to rank their average pain for the last 24 hours.
Change in Erectile function using the International Index of Erectile Function 5 (IIEF-5). | IIEF-5 will be assessed at baseline, and 1,3 and 6 months.
  Erectile function is estimated using the IIEF-5 which is a 5 item questionnaire. Based on the patients answers a final score is merged. The definition of erectile dysfunction(ED) is; 5-7 (severe), 8-11(moderate), 12-16(mild-moderate), 17-21(mild) and 22-25 no ED.
Change in Peyronies disease questionnaire score | Peyronies disease questionnaire will be assessed at baseline, and 1,3 and 6 months.
  Questionnaire to evaluate the psychological/physical consequences of peyronies disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense university hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided